CLINICAL TRIAL: NCT02050308
Title: Web-based Smoking Cessation Program for Tribal College Students
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Won Choi, PhD, MPH (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Won Choi, PhD, MPH, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13613; R01CA174481 (NIH)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Chewing Gum; Transdermal Patch; Bupropion; Varenicline; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-All Nations Breath of Life (I-ANBL) (Experimental): The culturally-tailored program includes 9 individual Internet-based sessions across a 12 week period and an additional individual Internet-based session at 6 months. Web sessions will last about half-an-hour (30 minutes) and will discuss topics that are important to quitting smoking (like: preparing to quit, dealing with cravings, and support systems, etc.) and topics relevant to American Indian culture (like traditional use of tobacco).
  We plan to give participants in our cessation program a choice of varenicline, bupropion, nicotine replacement therapy or no pharmacotherapy. We choose to give our participants a choice because our experience shows that we would be unlikely to recruit AI participants into a trial that requires pharmacotherapy use.
  Interventions: Other: Internet-All Nations Breath of Life (I-ANBL); Drug: Nicotine gum, Patch, or Lozenge or Zyban® or Chantix®
- Honoring the Gift of Heart Health (Active Comparator): The culturally-tailored program includes 9 individual Internet-based sessions across a 12 week period and an additional individual Internet-based session at 6 months. Web sessions will last about half-an-hour (30 minutes) and will discuss topics that are important to heart health (like: Assessing risk for heart disease, increasing fruit and vegetable consumption, physical activity, etc.).
  We plan to give participants in our cessation program a choice of varenicline, bupropion, nicotine replacement therapy or no pharmacotherapy. We choose to give our participants a choice because our experience shows that we would be unlikely to recruit AI participants into a trial that requires pharmacotherapy use.
  Interventions: Other: Honoring the Gift of Heart Health; Drug: Nicotine gum, Patch, or Lozenge or Zyban® or Chantix®

INTERVENTIONS:
Other: Internet-All Nations Breath of Life (I-ANBL) — * Participants will be asked to log into the website prior to the first session to allow for any problems with the site to be fixed prior to sessions starting. Topics we anticipate covering include, but are not limited to: preparing to quit, dealing with cravings, support systems, traditional tobacco, stress reduction, weight management, and staying quit, along with other topics determined during program development. For each session, the tribal college student will begin the session by answering a series of questions to produce an individually-tailored report that will be provided on the screen at the end of each week's session so that the smoker can work on strategies during the week before the next internet session
  * Weekly procedures will follow the same format as for the first session
  Arms: Internet-All Nations Breath of Life (I-ANBL)
Other: Honoring the Gift of Heart Health — These sessions help American Indians learn about what they can do to prevent heart disease. We will emphasize the increase consumption of fruits and vegetables as well as addressing other heart healthy activities. Honoring the Gift of Heart Health is a user-friendly program developed especially for American Indians. The manual provides the "how-to" for leading group education sessions. It offers "hands-on" activities that help people build the skills they need to make simple, practical, and lasting changes to help them fight heart disease. The protocol will follow procedures as the I-ANBL arm, however, this fruit and vegetable arm will not include individually tailored components, but just interactive web-based materials related to increasing heart health, including certain activities.
  Arms: Honoring the Gift of Heart Health
Drug: Nicotine gum, Patch, or Lozenge or Zyban® or Chantix® — Regardless of the intervention arm to which subjects are assigned, they will choose the option of nicotine replacement therapy they want, as long as they are eligible for it. All participants are offered the medications, but they do not have to take any medication to participate in the study.
  Other Names: Nictotine Replacement Therapy (Nicotine gum, Patch, or Lozenge) or Pharmacotherapy (Zyban® or Chantix®)

SUMMARY:
The purpose of this study is to test the effectiveness of a culturally-tailored Internet-based program that helps American Indian (AI) tribal college students quit smoking.

DETAILED DESCRIPTION:
Many of the approximately 25,000 American Indian (AI) students enrolled in tribal colleges/universities in the US arrive there as smokers. A 2011 study of high school seniors reported that the smoking prevalence among AI students is approximately 40%, the highest rate among all racial and ethnic groups studied. Although prevalence data on smoking among AI college students are limited, studies have shown that the majority of smokers in high school continue to smoke once they reach college. Prohibited from marketing to adolescents and children, the tobacco industry in recent years has shifted its most intense marketing to college students, resulting in increases in smoking rates among them. The transition to college provides amble opportunities for young adults to acquire new and harmful habits. Many of these habits do not seem so alien to young AIs: Cigarette smoking is the number one cause of preventable death among AIs. Cancer is the second leading cause of death among AIs, and lung cancer is the leading cause of cancer deaths for both AI men and women. Cultural factors, socioeconomic circumstances, and lack of culturally-tailored cessation programs for American Indian tribal college students have prevented access to effective interventions that promote smoking cessation. To date, few studies have focused on methods to encourage smoking cessation among tribal college students and no randomized clinical trials have yet been conducted. To address this public health deficit, we propose an innovative, effective, culturally and individually-tailored smoking cessation programs to promote cessation.

Primary aim is to: To test the effectiveness of a culturally-tailored internet-based smoking cessation intervention (I-ANBL) compared to an internet-based heart healthy diet (I-FV:fruit/vegetable) control condition in a randomized controlled trial with Tribal College students. Our hypothesis is that American Indian tribal college students randomized to the culturally-tailored smoking cessation arm will have significantly higher 7-day point prevalence abstinence (defined as no cigarettes in the past 7 days, biochemically verified) rates at 6 months than those receiving the heart healthy diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled at Salish Kootenai College
* Have a valid telephone number and email address
* Willing to participate in all study components
* Willing to be followed-up for 6 months
* Self identifies as American Indian or Alaska Native
* Is a current smoker

Exclusion Criteria:

* Planning to leave college within next 6 months
* Medically ineligible as a result of screening questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2015-05; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won Choi, PhD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Salish Kootenai College, Pablo, Montana

RESULTS

PARTICIPANT FLOW:
Groups:
- Honoring the Gift of Heart Health: The culturally-tailored program includes 9 individual Internet-based sessions across a 12 week period and an additional individual Internet-based session at 6 months. Web sessions will last about half-an-hour (30 minutes) and will discuss topics that are important to heart health (like: Assessing risk for heart disease, increasing fruit and vegetable consumption, physical activity, etc.).
  Participants in our cessation program have a choice of varenicline, bupropion, nicotine replacement therapy or no pharmacotherapy.
- Internet-All Nations Breath of Life (I-ANBL): The culturally-tailored program includes 9 individual Internet-based sessions across a 12 week period and an additional individual Internet-based session at 6 months. Web sessions will last about half-an-hour (30 minutes) and will discuss topics that are important to quitting smoking (like: preparing to quit, dealing with cravings, and support systems, etc.) and topics relevant to American Indian culture (like traditional use of tobacco).
  Participants in our cessation program have a choice of varenicline, bupropion, nicotine replacement therapy or no pharmacotherapy.
Period: Overall Study
Arm/Group | Honoring the Gift of Heart Health | Internet-All Nations Breath of Life (I-ANBL)
Started | 127 | 124
Completed | 28 | 22
Not Completed | 99 | 102

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Honoring the Gift of Heart Health | Internet-All Nations Breath of Life (I-ANBL) | Total
Number analyzed (Participants) | 127 | 124 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 127 | 124 | 251
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The row populations only includes participants with available data.
  Participants
    number analyzed (Participants) | 126 | 124 | 250
    Female | 67 | 61 | 128
    Male | 59 | 63 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 127 | 124 | 251
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 127 | 124 | 251

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 7-day Point Prevalence Abstinence
Description: self-reported and biochemically (salivary cotinine) verified point prevalence abstinence, defined as no smoking for the previous 7 days, at the 6-month follow-up.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Honoring the Gift of Heart Health | Internet-All Nations Breath of Life (I-ANBL)
Number analyzed (Participants) | 127 | 124
Participants | 9 | 9

2. Secondary Outcome: Cigarettes Per Day
Description: effect of intervention on the number of cigarettes smoked daily among those who continue to smoke at Month 6
Time Frame: Change from Baseline in number of cigarettes smoked daily at 6 months
Population: Smokers who were randomized to the Internet All Nations Breath of Life intervention or the Heart Healthy arm focusing on increasing fruits and vegetables.
  Due to very low retention rate at 6 months (less than 20%), no data were collected at 6 months.
  Therefore, the data below are baseline mean number of cigarettes smoked by intervention arm.
Measure: Mean (Standard Deviation); unit: Cigarettes/day
Groups:
- Internet All Nations Breath of Life: Internet based All Nations Breath of Life Smoking Cessation program
- Honoring the Gift of Heart Health: Internet based heart healthy program to increase fruits and vegetables
Arm/Group | Internet All Nations Breath of Life | Honoring the Gift of Heart Health
Number analyzed (Participants) | 124 | 127
Cigarettes/day | 4.00 (5.15) | 5.43 (5.42)

3. Secondary Outcome: Number of Quit Attempts
Description: comparison of the number of serious quit attempts between the two groups using Poisson regression
Time Frame: 6 months
Population: Overall retention at 6 months was low at 20% so no data were collected at 6 months.
Groups:
- I-ANBL: Internet All Nations Breath of Life
- Honoring the Gift of Heart Health: Increasing fruit and vegetable consumption
Arm/Group | I-ANBL | Honoring the Gift of Heart Health
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants Who Participated in All Sessions Over the Course of 6 Months.
Description: Number of participants who participated in all online sessions and study protocol procedures over the course of 6 months
Time Frame: 6 months
Population: The overall retention rate at 6 months was low at 20% so no data were collected at 6 months.
Arm/Group | Internet All Nations Breath of Life | Honoring the Gift of Heart Health
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Honoring the Gift of Heart Health | Internet-All Nations Breath of Life (I-ANBL)
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/124
Other Adverse Events (participants affected / at risk) | 0/127 | 0/124

LIMITATIONS AND CAVEATS:
Significant loss to follow-up, lower than expected salivary collection rates, and lower long-term retention of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT02050308/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT02050308/SAP_001.pdf